CLINICAL TRIAL: NCT06568367
Title: A Multi-center, Randomized, Double-blind, Placebo-controlled Trial to Assess the Efficacy and Safety of Solriamfetol in Excessive Sleepiness Associated With Shift Work Disorder
Brief Title: Studying Solriamfetol Modulation of TAAR-1, Dopamine, and Norepinephrine in Shift Work Disorder (SUSTAIN)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Axsome Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SOL-SWD-301
Record Dates: First submitted 2024-08-21; First posted 2024-08-23 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Excessive Sleepiness; Shift-work Disorder
Keywords: Excessive Sleepiness; Solriamfetol; Sunosi; SWD; Dopamine norepinephrine reuptake inhibitor; Non-stimulant therapy; Insomnia; Circadian Rhythm Sleep Disorder; Trace amine-associated receptor 1 (TAAR1) agonist
MeSH Terms: conditions — Disorders of Excessive Somnolence; Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm | interventions — solriamfetol

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Solriamfetol 150mg (Experimental): Up to 12 weeks
  Interventions: Drug: Solriamfetol 150 mg
- Solriamfetol 300mg (Experimental): Up to 12 weeks
  Interventions: Drug: Solriamfetol 300 mg
- Placebo (Placebo Comparator): Up to 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Solriamfetol 150 mg — Solriamfetol tablets, taken once daily
  Arms: Solriamfetol 150mg
Drug: Solriamfetol 300 mg — Solriamfetol tablets, taken once daily
  Arms: Solriamfetol 300mg
Drug: Placebo — Placebo tablets, taken once daily
  Arms: Placebo

SUMMARY:
SUSTAIN (Studying Solriamfetol Modulation of TAAR-1, Dopamine, and Norepinephrine in Shift Work Disorder) is a Phase 3, multi-center, randomized, double-blind, placebo-controlled, parallel- group trial to assess the efficacy and safety of solriamfetol in adults with excessive sleepiness associated with shift work disorder (SWD).

DETAILED DESCRIPTION:
Eligible subjects must meet the International Classification of Sleep Disorders, Third Edition (ICSD-3) criteria for Shift Work Disorder (SWD). Subjects will be randomized in a 1:1:1 ratio to receive solriamfetol titrated to either 150 mg, 300 mg, or placebo once per night shift for 12 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Meets International Classification of Sleep Disorders, Third Edition (ICSD-3) criteria for Shift Work Disorder (SWD)
* Provides written informed consent to participate in the study before the conduct of any study procedures.
* Male or female, aged 18 to 65 inclusive.

Exclusion Criteria:

* Prior exposure to solriamfetol/Sunosi, through either a clinical study or prescription.
* Unable to comply with study procedures.
* Medically inappropriate for study participation in the opinion of the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2024-08-01 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Change from Baseline to Week 12 in the mean sleep latency time as measured by the Maintenance of Wakefulness Test (MWT). | 12 weeks
Change from Baseline to Week 12 in the Clinical Global Impressions of Severity of Illness (CGI-S) for sleepiness during the night shift. | 12 weeks

CONTACTS AND LOCATIONS:
Locations (37):
- United States (35):
  - Clinical Research Site, Cullman, Alabama
  - Clinical Research Site, Chandler, Arizona
  - Clinical Research Site, Tucson, Arizona
  - Clinical Research Site, Little Rock, Arkansas
  - Clinical Research Site, Cerritos, California
  - Clinical Research Site, Chula Vista, California
  - Clinical Research Site, Huntington Beach, California
  - Clinical Research Site, Long Beach, California
  - Clinical Research Site, Santa Ana, California
  - Clinical Research Site, Colorado Springs, Colorado
  - Clinical Research Site, Brandon, Florida
  - Clinical Research Site, Hialeah, Florida
  - Clinical Research Site, Miami, Florida
  - Clinical Research Site, Miami Lakes, Florida
  - Clinical Research Site, Atlanta, Georgia
  - Clinical Research Site, Stockbridge, Georgia
  - Clinical Research Site, Towson, Maryland
  - Clinical Research Site, Boston, Massachusetts
  - Clinical Research Site, Lansing, Michigan
  - Clinical Research Site, Novi, Michigan
  - Clinical Research Site, Southfield, Michigan
  - Clinical Research Site, Chesterfield, Missouri
  - Clinical Research Site, St Louis, Missouri
  - Clinical Research Site, Henderson, Nevada
  - Clinical Research Site, Middletown, New Jersey
  - Clinical Research Site, Denver, North Carolina
  - Clinical Research Site, Fayetteville, North Carolina
  - Clinical Research Site, Huntersville, North Carolina
  - Clinical Research Site, Cincinnati, Ohio
  - Clinical Research Site, Wyomissing, Pennsylvania
  - Clinical Research Site, Charleston, South Carolina
  - Clinical Research Site, Columbia, South Carolina
  - Clinical Research Site, Houston, Texas
  - Clinical Research Site, San Antonio, Texas
  - Clinical Research Site, Sugar Land, Texas
- Canada (2):
  - Clinical Research Site, Markham, Ontario
  - Clinical Research Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: SUSTAIN Study Website — https://www.SustainSWD.com
- See also: Axsome Therapeutics Website — http://axsome.com